CLINICAL TRIAL: NCT02787512
Title: A Randomized Controlled Trial for Preoperative Biliary Drainage With Metal Versus Plastic Stents in Patients With Periampullary Cancer
Brief Title: Preoperative Biliary Drainage With Metal Versus Plastic Stents in Periampullary Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SNUBH-IMGPB-2016-01
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-10

CONDITIONS: Jaundice; Periampullary Cancer
Keywords: ERCP; stent; preoperative biliary drainage
MeSH Terms: conditions — Jaundice | interventions — Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plastic stent (Active Comparator): 10 Fr plastic stent (Percuflex Amsterdam® or C-flex pigtail® or Advanix® Biliary stent)
  Interventions: Device: Stent
- Uncovered metal stent (Experimental): Uncovered metal stent (WallFlex® Biliary RX stent)
  Interventions: Device: Stent

INTERVENTIONS:
Device: Stent — Endoscopic biliary stent insertion

SUMMARY:
Currently, routine preoperative biliary drainage (PBD) was not recommended. However, PBD is still necessary in case of patients with cholangitis or very high level of bilirubin or patients who are expected to receive delayed surgery.

The aim of this clinical trial is to demonstrate non-inferiority of uncovered self-expandable metal stent to plastic stent for PBD by endoscopic retrograde cholangiopancreatography in patients with periampullary cancer undergoing curative intent pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Jaundice is one of the most common symptoms in patients with periampullary cancers including pancreatic cancer, common bile duct (CBD) cancer, ampulla of Vater (AoV) cancer, and duodenal cancer. Traditionally, preoperative biliary drainage (PBD) was routinely performed in these cancers because it might favorably influence sepsis, endotoxemia, and intravascular coagulation. However, a recent randomized control study reported that routine PBD in patients undergoing surgery for cancer of the pancreatic head increases the rate of complications. Therefore, routine PBD was not recommended. However, PBD is still necessary in case of patients with cholangitis or very high level of bilirubin or patients who are expected to receive delayed surgery.

In these patients with necessity of PBD, a plastic stent (PS) has been used because it is good for temporary use with cheap prices. However, it is sometimes occluded before surgery or not enough for rapid decompressing jaundice mainly because of its short diameter. In this aspect, a self-expandable metal stent (SEMS) has strength compared to PS because it has a longer diameter which enables rapid decompression with a fewer events of occlusion. However, SEMS is much more expensive than PS and the exact length of stent is more critical.

Although there are still lack of evidence which compares the results between PS and SEMS, National Comprehensive Cancer Network (NCCN) guidelines recently recommended the use of a short SEMS for pancreatic adenocarcinoma patients with cholangitis or fever. However, we needed more concrete evidence about this principle.

ELIGIBILITY:
Inclusion Criteria:

A. Patients 20-80 years old B. Patients with surgically resectable periampullary cancer on CT scans with or without MRI or PET-CT scans C. ECOG Performance score 0 or 1 D. Patients who need preoperative biliary drainage (PBD) because of one or more of following causes

* Cholangitis defined as revised Tokyo guidelines
* Level of total bilirubin >= 10mg/dL
* Expected time to operation >= 7 days

Exclusion Criteria:

A. Patients who received previous endoscopic biliary drainage or percutaneous biliary drainage B. Patients with acute pancreatitis before PBD

C. Patients with bleeding tendency or coagulopathy or anticoagulation therapy as follows:

* Patients who take clopidogrel within 5 days before PBD
* Patients who take warfarin within 2 days before PBD
* Patients who receive heparin within 1 days before PBD D. Patients with pregnancy or suspected pregnancy E. Patients who are currently enrolled in another investigational trials that would directly interfere with current study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Reintervention rate until operation | Between preoperative biliary drainage and surgery
  Between preoperative biliary drainage and surgery, reintervention (re-preoperative biliary drainage) would be checked and analyzed.

SECONDARY OUTCOMES:
Other complication rate associated with endoscopic stent insertion and stent indwell | Between preoperative biliary drainage and surgery
  Until surgery, preoperative biliary drainage associated with complication would be checked and analyzed.
Rate of decrease of total bilirubin | Between preoperative biliary drainage and surgery
  Amount of decrease of total bilirubin between preoperative biliary drainage and surgery would be checked.
Time to operation | Between preoperative biliary drainage and surgery
  Interval between preoperative biliary drainage and surgery would be checked.
Time to hospital discharge after pancreaticoduodenectomy | 6 month
  Interval between surgery and discharge would be checked.
Mortality until 3 months after pancreaticoduodenectomy | 3 month
  The mortality rate would be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Jaihwan Kim, MD, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Gaag NA, Rauws EA, van Eijck CH, Bruno MJ, van der Harst E, Kubben FJ, Gerritsen JJ, Greve JW, Gerhards MF, de Hingh IH, Klinkenbijl JH, Nio CY, de Castro SM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for cancer of the head of the pancreas. N Engl J Med. 2010 Jan 14;362(2):129-37. doi: 10.1056/NEJMoa0903230. PMID 20071702
- [Background] Adams MA, Anderson MA, Myles JD, Khalatbari S, Scheiman JM. Self-expanding metal stents (SEMS) provide superior outcomes compared to plastic stents for pancreatic cancer patients undergoing neoadjuvant therapy. J Gastrointest Oncol. 2012 Dec;3(4):309-13. doi: 10.3978/j.issn.2078-6891.2011.050. PMID 23205306
- [Background] Decker C, Christein JD, Phadnis MA, Wilcox CM, Varadarajulu S. Biliary metal stents are superior to plastic stents for preoperative biliary decompression in pancreatic cancer. Surg Endosc. 2011 Jul;25(7):2364-7. doi: 10.1007/s00464-010-1552-6. Epub 2011 Mar 4. PMID 21373939